CLINICAL TRIAL: NCT06758271
Title: Special Drug Use-results Survey for Long-term Use
Brief Title: Special Drug Use-results Survey for Long-term Use（Avacopan）
Status: Recruiting | Type: Observational
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TVPMS01
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Microscopic Polyangiitis (MPA); Granulomatosis With Polyangiitis (GPA)
MeSH Terms: conditions — Microscopic Polyangiitis; Granulomatosis with Polyangiitis | interventions — avacopan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Avacopan treatmented
  Interventions: Drug: Avacopan

INTERVENTIONS:
Drug: Avacopan — oral administration

SUMMARY:
The purpose of this survey is evaluating the safety and efficacy of long-term administration of avacopan for Japanese patients with microscopic polyangiitis or granulomatosis with polyangiitis under actual conditions of use.

DETAILED DESCRIPTION:
The purpose of this survey is evaluating the safety and efficacy of long-term administration of avacopan for Japanese patients with microscopic polyangiitis or granulomatosis with polyangiitis under actual conditions of use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with granulomatosis with polyangiitis or microscopic polyangiitis who are treatment with avacopan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with granulomatosis with polyangiitis or microscopic polyangiitis who are treatment with avacopan
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Research site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No